CLINICAL TRIAL: NCT05674994
Title: Glucocorticoids Versus Placebo for the Treatment of Acute Exacerbation of Idiopathic Pulmonary Fibrosis: a Randomized Controlled Trial
Brief Title: Glucocorticoids Versus Placebo for the Treatment of Acute Exacerbation of Idiopathic Pulmonary Fibrosis
Acronym: EXAFIP2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EXAFIP2
Record Dates: First submitted 2022-12-09; First posted 2023-01-09 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Acute Exacerbation of Idiopathic Pulmonary Fibrosis
MeSH Terms: interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MethylPrednisone/Prednisone (Experimental): * Day 1, 2 and 3: Intravenous Methylprednisolone 10 mg/kg/d (without exceeding 1000 mg/d) Vials of injectable solution of methylprednisolone® are diluted in 100 ml of NaCl 0.9% or G5%. Perfusion duration is between 20 to 30 minutes. The commercialized form for methylprednisolone injectable solution is not imposed and is taken from the stock of each pharmacy of the participating centers.
  * From day 4 to Day 30: Oral Prednisone slow tappering
    * 1 mg/kg/d for 7 days
    * 0.5 mg/kg/d for 7 days
    * 0.25 mg/kg/d for 7 days,
    * 10 mg/d until Day 30. For 10mg/kg, 1 mg/kg, 0.5 mg/kg, 0.25 mg/kg; rounding to 5 decimal lower if decimal ≤ 7 and the top ten if decimal ≥ 8.
  Interventions: Drug: Methylprednisone/Prednisone
- Placebo (Placebo Comparator): * Day 1, 2 and 3: Intravenous Methylprednisolone-Placebo
  * From Day 4 to Day 30: Oral Prednisone-Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Methylprednisone/Prednisone — Patients will be enrolled during their hospitalization in pneumology department, as part of current practice, within 7 days of the screening visit. The investigator will perform randomization by connecting to the eCRF, randomization be stratified for the severity of IPF and the treatment with antifibrotic therapy (Nintedanib or Pirfenidone) (yes/no).
  If patient is randomized in Glucocorticoids Group:
  * Day 1, 2 and 3: Intravenous Methylprednisolone 10 mg/kg/d (without exceeding 1000 mg/d). Vials of injectable solution of methylprednisolone® are diluted in 100 ml of NaCl 0.9% or G5%. Perfusion duration is between 20 to 30 minutes.
  * From day 4 to Day 30: Oral Prednisone slow tappering
    * 1 mg/kg/d for 7 days
    * 0.5 mg/kg/d for 7 days
    * 0.25 mg/kg/d for 7 days,
    * 10 mg/d until Day 30. For 10mg/kg, 1 mg/kg, 0.5 mg/kg, 0.25 mg/kg; rounding to 5 decimal lower if decimal ≤ 7 and the top ten if decimal ≥ 8.
  Arms: MethylPrednisone/Prednisone
Other: Placebo — Patients will be enrolled during their hospitalization in pneumology department, as part of current practice, within 7 days of the screening visit. The investigator will perform randomization by connecting to the eCRF, randomization be stratified for the severity of IPF and the treatment with antifibrotic therapy (Nintedanib or Pirfenidone) (yes/no).
  If patient is randomized in Placebo Group:
  Day 1, 2 and 3: Intravenous Methylprednisolone-Placebo From Day 4 to Day 30: Oral Prednisone-Placebo The Methylprednisolone-Placebo corresponds to 100 ml of NaCl 0.9 % or G5%. Perfusion duration is between 20 to 30 minutes.
  For the Prednisone-Placebo, the placebo was an oral solution formulated with a bittering agent (pharmaceutical excipient). Specifically, in place of prednisone, sucrose octaacetate (defined as a GRAS-'Generally Recognized as Safe' excipient by the EMA) was used at 5 mg/mL.
  Arms: Placebo

SUMMARY:
Acute exacerbation of idiopathic pulmonary fibrosis (AE-IPF) is associated with a poor prognosis, with a 3-month mortality rate of over 50%. To date, no treatment has been proven to be effective in AI-FPI. The interest of glucocorticoids is controversial and needs to be confirmed. This confirmation is mandatory to validate the improvement of the prognosis of EA-IPF under this treatment but also to search for unsuspected deleterious effects as it has been shown with immunosuppressants in stable idiopathic pulmonary fibrosis.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is the most frequent idiopathic interstitial lung disease (ILD) in adults. Its prognosis is poor with a median survival time ranging from 2 to 3 years. Acute exacerbation of IPF (IPF-AE) is defined as acute, clinically significant respiratory deterioration characterized by evidence of new widespread alveolar abnormalities. Recently, diagnosis criteria were defined now allowing standardized diagnosis of IPF-AE and thus its study. IPF-AE is a major event of the disease having a 5 to 10% annual incidence. In-hospital mortality after IPF-AE exceeds 50% and current evidence suggests that up to 46% of deaths in IPF patients are associated with IPF-AE.

For the time being, no treatment has been proved to be effective in IPF-AE. While the clinical practice guideline suggests treatment with steroids, this recommendation is based only on expert opinion (low level evidence). Retrospective studies suggested the efficacy of thrombomodulin, cyclophosphamide or of therapeutic strategy including plasma exchange, rituximab and intravenous immunoglobulins. A recent Japanese randomized trial failed to show the efficacy of thrombomodulin alfa. Investigators performed a randomized trial assessing the role of cyclophosphamide on top of pulse steroid (EXAFIP-NCT02460588) and showed that cyclophosphamide did not reduce the 3-month mortality. A study assessing the effect of therapeutic plasma exchange, rituximab and intravenous immunoglobulins for severe form of IPF-AE patients admitted to Intensive Care Unit (ICU) is still ongoing (NCT03286556). Presently, the clinical benefit of corticosteroids is questioned. Indeed, 2 retrospective series reported an absence of outcome improvement by corticosteroids among IPF-AE patients and even suggested a potential detrimental outcome.

It is therefore necessary to set-up a placebo-controlled randomized trial: investigator's goal is to test the hypothesis that a corticosteroid treatment is highly efficient in IPF-AE, compared to placebo.

This underlines that, as no good evidence is available to support the use of glucocorticoids in IPF-AE, randomized controlled trials are also needed to address their efficacy and safety in this indication.

The choices of glucocorticoids' dosage, primary objective (mortality) and primary assessment criteria (all cause mortality rate at Day 30) are driven by investigator's previous study, EXAFIP. In this study, glucocorticoids dosage was as follow: intravenous methylprednisolone, 10 mg/kg/d (without exceeding 1000 mg/d), 3 days in a row shift to prednisone at 1 mg/kg/d for 1 week, and 0.75 mg/kg/d for 1 week, then 0.5 mg/kg/d for 1 week, and 0.25 mg/kg/d for 1 week, and 10 mg/d if weight > 65 kg; 7.5 mg if weight ≤ 65 kg until M6. The 1-month mortality of patient under this high dose of glucocorticoids was 20%.

In view of the poor prognosis of IPF-AE, it seems also important to evaluate the effect of treatment on overall mortality at Day 90.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 years of age
2. IPF or IPF (likely) diagnosis defined on 2018 international recommendations
3. Definite or suspected Acute Exacerbation defined by the international working group criteria after exclusion of alternative diagnoses of acute worsening

   *The criteria of IPF-AE are as follows:
   * Previous or concurrent diagnosis of IPF (a)
   * Acute worsening or development of dyspnea typically < 1-month duration
   * Computed tomography with new bilateral ground-glass opacity and/or consolidation superimposed on a background pattern consistent with usual interstitial pneumonia pattern (b)
   * Deterioration not fully explained by cardiac failure or fluid overload Patients who fail to meet all 4 criteria due to missing computed tomography should be considered as having "suspected Acute Exacerbation".

     1. If the diagnosis of IPF is not previously established, this criterion can be met by the presence of radiologic and/or histopathologic changes consistent with usual interstitial pneumonia pattern on the current evaluation.
     2. If no previous computed tomography is available, the qualifier "new" can be dropped from the third criterion.
4. For women of childbearing age: efficient contraception for the duration of the study*

   *Effective contraception is defined as any contraceptive method that is used consistently and appropriately and has a low failure rate (i.e., less than 1% per year)
5. Affiliation to the social security
6. Patient able to understand and sign a written informed consent form or in case of incapacity of the patient to a relative whom understand and sign a written informed consent form

Exclusion Criteria:

1. Identified etiology for acute worsening (i.e.: infectious disease)
2. Known hypersensitivity to glucocorticoids or to any component of the study treatment
3. Patient requiring mechanical ventilation or already on mechanical ventilation
4. Active bacterial, viral, fungal or parasitic infection. On swab collected, only positive for SARS-CoV-2, Influenzae A, Influenzae B and Respiratory Syncytial Virus (RSV) result, are considered active viral infection. The others viruses (i.e. Rhinovirus, Adenovirus…) are not considered to be responsible of pneumonia.
5. Active cancer
6. Patient on a lung transplantation waiting list
7. Treatment with glucocorticoids > 1 mg/kg/d from more than 7 days in the last 15 days
8. Patient participating to another interventional clinical trial
9. Documented pregnancy or lactation
10. Patient under tutorship or curatorship
11. Patient deprived of liberty
12. Patient under court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2025-10-25 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of glucocorticoids compared to placebo on mortality | Day 30
  This outcome corresponds to the all-cause mortality rate at day 30.

SECONDARY OUTCOMES:
Time to death at Day 30 | Day 30
  This outcome corresponds to the vital status assessment at Day 30 with time (in days) between randomization and death.
Time to death at Day 90 | Day 90
  This outcome corresponds to the vital status assessment at Day 90 with time (in days) between randomization and death.
Death or transplantation at Day 90 | Day90
  This outcome corresponds to the vital status and transplantation at Day 90.
Respiratory disease-specific mortality rate at Day 30 | Day 30
  This outcome corresponds to the mortality linked to the respiratory disease: cause of death assessment at Day 30.
Respiratory disease-specific mortality rate at Day 90 | Day 90
  This outcome corresponds to the mortality linked to the respiratory disease: cause of death assessment at Day 90.
Time to worsening | Day30
  This outcome corresponds to the time (in days) from randomization to worsening from day4 to day30 (end of study treatment).
Percentage of patients admitted to ICU | Day90
  This outcome corresponds to the percentage of patients admitted to ICU from randomization to ICU's admission.
Percentage of patients requiring invasive ventilation | Day90
  This outcome corresponds to the percentage of patients requiring invasive ventilation from randomization to invasive ventilation.
Length of hospital stay | Day 90
  This outcome corresponds to the length of hospital-stay: Time (in days) from randomization to hospital withdraw.
Radiological evolution | Day90
  This outcome corresponds to the progression of pulmonary fibrosis: Chest HRCT scan comparison before Acute Exacerbation (if available) and at Day 90. Chest CT scans exacerbation, were analyzed by 2 thoracic radiologists' expert in interstitial lung diseases (PYBrillet, MPDebray). Before chest CT scans were evaluated for the pattern of ILD, according to the 2018 ATS/ERS classification for the diagnosis of IPF. The extent of interstitial fibrosing features on "Before" and "D90" CT scan was calculated by summing the extent of honeycombing, the extent of ground glass attenuation causing traction bronchiectasis both to the nearest 5% of the whole lungs, and the extent of reticular opacities. For this latter, the extension was estimated to the nearest 10% at three lung zones (delimited by the carina and the lowest inferior pulmonary vein for both lungs) and averaged between these 3 zones.
Pulmonary function tests evolution: Forced Vital Capacity | Day90
  This outcome corresponds to the Absolute change in percent Forced Vital Capacity: Pulmonary function tests (PFTs) comparison before Acute Exacerbation (if available) and at Day 90.
Pulmonary function tests evolution: DLCO | Day90
  This outcome corresponds to the Absolute change in percent DLCO: Pulmonary function tests (PFTs) comparison before Acute Exacerbation (if available) and at Day 90.
Occurence of Infectious disease | Day 90
  This outcome corresponds to the occurence of infectious disease from D1 to Day 90.
Occurence of Diabetes mellitus | Day90
  This outcome corresponds to the occurence of diabetes mellitus by Capillary blood glucose monitoring and/or fasting blood glucose daily from D1 to Day 90.
Occurence of Cardiovascular disorder | Day90
  This outcome corresponds to the occurence of cardiovascular disorder (heart rate, blood pressure, clinical history daily) from D1 to Day 90.
Occurence of Neuropsychological disturbances | Day90
  This outcome corresponds to the occurence of neuropsychological disturbances from D1 to Day 90.
Occurence of Clinical laboratory evaluation | Day 90
  This outcome corresponds to the occurence of clinical laboratory evolution (blood count, serum chemistries and creatinin measurement) from Day 4 to Day 90.
Compare both arms in terms of Dyspnea | Day1, Day30, Day90
  This outcome corresponds to the 0-100-mm visual analogue (VAS) scale anchored with 0 ''no breathlessness'' and 10 or 100 ''worst imaginable breathlessness", at Day1, Day 30 and Day 90.
Compare both arms in terms of Anxiety | Day 90
  This outcome corresponds to theHospital Anxiety and Depression Scale (HADs), daily from randomization to hospital withdraw, Day 30 and Day 90. The HAD scale is an instrument that screens for anxiety and depressive disorders. It includes 14 questions rated from 0 to 3. Seven questions relate to anxiety (Total A) and seven others to the depressive dimension (Total D), thus making it possible to obtain both scores (maximum score for each score = 21).
Compare both arms in terms of Depression | Day90
  This outcome corresponds to the Anxiety and Depression Scale (HADs), from Day 1 to Day 90. The HAD scale is an instrument that screens for anxiety and depressive disorders. It includes 14 questions rated from 0 to 3. Seven questions relate to anxiety (Total A) and seven others to the depressive dimension (Total D), thus making it possible to obtain both scores (maximum score for each score = 21).
Compare both arms in terms of Clinical status at day 15 | Day15
  This outcome corresponds to the -category ordinal scale: 1: not hospitalized and no limitations of activities, 2: not hospitalized, with limitations of activities, home oxygen requirement, or both, 3: hospitalized, not requiring supplemental oxygen and no longer requiring ongoing medical care (used if hospitalization was extended for infection-control or other nonmedicala reason, 4: hospitalized requiring any supplemental oxygen, 5: hospitalized, requiring use of high high-flow oxygen device or noninvasive ventilation, 6: hospitalize, receiving invasive mechanicalventilation or extra corporeal membrane oxygenation (ECMO), 7: death.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc NACCACHE, Study Director — Fondation Hôpital Saint-Joseph
Locations (29):
- France (29):
  - CHU ANgers, Angers
  - CHU de Besancon, Besançon
  - Hôpital Avicenne, Bobigny
  - CHU BOrdeaux, Bordeaux
  - CHU Caen, Caen
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHIC, Créteil
  - CHU de Dijon, Dijon
  - CHU Grenoble, Grenoble
  - CHRU Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - Hôpital Nord, Marseille
  - CHU de Montpellier, Montpellier
  - CHU Nancy, Nancy
  - CHU de Nantes, Nantes
  - CHU Nice, Nice
  - Hôpital Paris Saint-Joseph, Paris
  - Hôpital Bichat, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital FOCH, Paris
  - Hôpital Kremiln Bicetre, Paris
  - Hôpital Saint-Louis, Paris
  - Hôpital Tenon, Paris
  - CHU Reims, Reims
  - CHU Rennes, Rennes
  - CHU Rouen, Rouen
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours

REFERENCES:
- [Background] Naccache JM, Montil M, Cadranel J, Cachanado M, Cottin V, Crestani B, Valeyre D, Wallaert B, Simon T, Nunes H. Study protocol: exploring the efficacy of cyclophosphamide added to corticosteroids for treating acute exacerbation of idiopathic pulmonary fibrosis; a randomized double-blind, placebo-controlled, multi-center phase III trial (EXAFIP). BMC Pulm Med. 2019 Apr 11;19(1):75. doi: 10.1186/s12890-019-0830-x. PMID 30971235
- [Background] Naccache JM, Jouneau S, Didier M, Borie R, Cachanado M, Bourdin A, Reynaud-Gaubert M, Bonniaud P, Israel-Biet D, Prevot G, Hirschi S, Lebargy F, Marchand-Adam S, Bautin N, Traclet J, Gomez E, Leroy S, Gagnadoux F, Riviere F, Bergot E, Gondouin A, Blanchard E, Parrot A, Blanc FX, Chabrol A, Dominique S, Gibelin A, Tazi A, Berard L, Brillet PY, Debray MP, Rousseau A, Kerjouan M, Freynet O, Dombret MC, Gamez AS, Nieves A, Beltramo G, Pastre J, Le Borgne-Krams A, Degot T, Launois C, Plantier L, Wemeau-Stervinou L, Cadranel J, Chenivesse C, Valeyre D, Crestani B, Cottin V, Simon T, Nunes H; EXAFIP investigators and the OrphaLung network. Cyclophosphamide added to glucocorticoids in acute exacerbation of idiopathic pulmonary fibrosis (EXAFIP): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Respir Med. 2022 Jan;10(1):26-34. doi: 10.1016/S2213-2600(21)00354-4. Epub 2021 Sep 7. PMID 34506761
- [Background] Raghu G, Remy-Jardin M, Myers JL, Richeldi L, Ryerson CJ, Lederer DJ, Behr J, Cottin V, Danoff SK, Morell F, Flaherty KR, Wells A, Martinez FJ, Azuma A, Bice TJ, Bouros D, Brown KK, Collard HR, Duggal A, Galvin L, Inoue Y, Jenkins RG, Johkoh T, Kazerooni EA, Kitaichi M, Knight SL, Mansour G, Nicholson AG, Pipavath SNJ, Buendia-Roldan I, Selman M, Travis WD, Walsh S, Wilson KC; American Thoracic Society, European Respiratory Society, Japanese Respiratory Society, and Latin American Thoracic Society. Diagnosis of Idiopathic Pulmonary Fibrosis. An Official ATS/ERS/JRS/ALAT Clinical Practice Guideline. Am J Respir Crit Care Med. 2018 Sep 1;198(5):e44-e68. doi: 10.1164/rccm.201807-1255ST. PMID 30168753
- [Background] Collard HR, Ryerson CJ, Corte TJ, Jenkins G, Kondoh Y, Lederer DJ, Lee JS, Maher TM, Wells AU, Antoniou KM, Behr J, Brown KK, Cottin V, Flaherty KR, Fukuoka J, Hansell DM, Johkoh T, Kaminski N, Kim DS, Kolb M, Lynch DA, Myers JL, Raghu G, Richeldi L, Taniguchi H, Martinez FJ. Acute Exacerbation of Idiopathic Pulmonary Fibrosis. An International Working Group Report. Am J Respir Crit Care Med. 2016 Aug 1;194(3):265-75. doi: 10.1164/rccm.201604-0801CI. PMID 27299520
- [Background] Kondoh Y, Azuma A, Inoue Y, Ogura T, Sakamoto S, Tsushima K, Johkoh T, Fujimoto K, Ichikado K, Matsuzawa Y, Saito T, Kishi K, Tomii K, Sakamoto N, Aoshima M, Araya J, Izumi S, Arita M, Abe M, Yamauchi H, Shindoh J, Suda T, Okamoto M, Ebina M, Yamada Y, Tohda Y, Kawamura T, Taguchi Y, Ishii H, Hashimoto N, Abe S, Taniguchi H, Tagawa J, Bessho K, Yamamori N, Homma S. Thrombomodulin Alfa for Acute Exacerbation of Idiopathic Pulmonary Fibrosis. A Randomized, Double-Blind Placebo-controlled Trial. Am J Respir Crit Care Med. 2020 May 1;201(9):1110-1119. doi: 10.1164/rccm.201909-1818OC. PMID 31917621
- [Background] Papiris SA, Kagouridis K, Kolilekas L, Papaioannou AI, Roussou A, Triantafillidou C, Baou K, Malagari K, Argentos S, Kotanidou A, Karakatsani A, Manali ED. Survival in Idiopathic pulmonary fibrosis acute exacerbations: the non-steroid approach. BMC Pulm Med. 2015 Dec 14;15:162. doi: 10.1186/s12890-015-0146-4. PMID 26666385
- [Background] Farrand E, Vittinghoff E, Ley B, Butte AJ, Collard HR. Corticosteroid use is not associated with improved outcomes in acute exacerbation of IPF. Respirology. 2020 Jun;25(6):629-635. doi: 10.1111/resp.13753. Epub 2019 Dec 17. PMID 31846126
- [Background] Nalysnyk L, Cid-Ruzafa J, Rotella P, Esser D. Incidence and prevalence of idiopathic pulmonary fibrosis: review of the literature. Eur Respir Rev. 2012 Dec 1;21(126):355-61. doi: 10.1183/09059180.00002512. PMID 23204124
- [Background] Duchemann B, Annesi-Maesano I, Jacobe de Naurois C, Sanyal S, Brillet PY, Brauner M, Kambouchner M, Huynh S, Naccache JM, Borie R, Piquet J, Mekinian A, Virally J, Uzunhan Y, Cadranel J, Crestani B, Fain O, Lhote F, Dhote R, Saidenberg-Kermanac'h N, Rosental PA, Valeyre D, Nunes H. Prevalence and incidence of interstitial lung diseases in a multi-ethnic county of Greater Paris. Eur Respir J. 2017 Aug 3;50(2):1602419. doi: 10.1183/13993003.02419-2016. Print 2017 Aug. PMID 28775045
- [Background] Cottin V, Crestani B, Cadranel J, Cordier JF, Marchand-Adam S, Prevot G, Wallaert B, Bergot E, Camus P, Dalphin JC, Dromer C, Gomez E, Israel-Biet D, Jouneau S, Kessler R, Marquette CH, Reynaud-Gaubert M, Aguilaniu B, Bonnet D, Carre P, Danel C, Faivre JB, Ferretti G, Just N, Lebargy F, Philippe B, Terrioux P, Thivolet-Bejui F, Trumbic B, Valeyre D. French practical guidelines for the diagnosis and management of idiopathic pulmonary fibrosis - 2017 update. Full-length version. Rev Mal Respir. 2017 Oct;34(8):900-968. doi: 10.1016/j.rmr.2017.07.017. Epub 2017 Sep 20. No abstract available. PMID 28939155
- [Background] Idiopathic Pulmonary Fibrosis Clinical Research Network; Raghu G, Anstrom KJ, King TE Jr, Lasky JA, Martinez FJ. Prednisone, azathioprine, and N-acetylcysteine for pulmonary fibrosis. N Engl J Med. 2012 May 24;366(21):1968-77. doi: 10.1056/NEJMoa1113354. Epub 2012 May 20. PMID 22607134
- [Background] Collard HR, Moore BB, Flaherty KR, Brown KK, Kaner RJ, King TE Jr, Lasky JA, Loyd JE, Noth I, Olman MA, Raghu G, Roman J, Ryu JH, Zisman DA, Hunninghake GW, Colby TV, Egan JJ, Hansell DM, Johkoh T, Kaminski N, Kim DS, Kondoh Y, Lynch DA, Muller-Quernheim J, Myers JL, Nicholson AG, Selman M, Toews GB, Wells AU, Martinez FJ; Idiopathic Pulmonary Fibrosis Clinical Research Network Investigators. Acute exacerbations of idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2007 Oct 1;176(7):636-43. doi: 10.1164/rccm.200703-463PP. Epub 2007 Jun 21. PMID 17585107
- [Background] Collard HR, Yow E, Richeldi L, Anstrom KJ, Glazer C; IPFnet investigators. Suspected acute exacerbation of idiopathic pulmonary fibrosis as an outcome measure in clinical trials. Respir Res. 2013 Jul 13;14(1):73. doi: 10.1186/1465-9921-14-73. PMID 23848435
- [Background] Churg A, Muller NL, Silva CI, Wright JL. Acute exacerbation (acute lung injury of unknown cause) in UIP and other forms of fibrotic interstitial pneumonias. Am J Surg Pathol. 2007 Feb;31(2):277-84. doi: 10.1097/01.pas.0000213341.70852.9d. PMID 17255773
- [Background] Parambil JG, Myers JL, Ryu JH. Histopathologic features and outcome of patients with acute exacerbation of idiopathic pulmonary fibrosis undergoing surgical lung biopsy. Chest. 2005 Nov;128(5):3310-5. doi: 10.1378/chest.128.5.3310. PMID 16304277
- [Background] Oda K, Ishimoto H, Yamada S, Kushima H, Ishii H, Imanaga T, Harada T, Ishimatsu Y, Matsumoto N, Naito K, Yatera K, Nakazato M, Kadota J, Watanabe K, Kohno S, Mukae H. Autopsy analyses in acute exacerbation of idiopathic pulmonary fibrosis. Respir Res. 2014 Sep 1;15(1):109. doi: 10.1186/s12931-014-0109-y. PMID 25176016
- [Background] Dotan Y, Vaidy A, Shapiro WB, Zhao H, Dass C, Toyoda Y, Marchetti N, Shenoy K, Cordova FC, Criner GJ, Mamary AJ. Effect of Acute Exacerbation of Idiopathic Pulmonary Fibrosis on Lung Transplantation Outcome. Chest. 2018 Oct;154(4):818-826. doi: 10.1016/j.chest.2018.06.027. Epub 2018 Jun 30. PMID 29966665
- [Background] Raghu G, Collard HR, Egan JJ, Martinez FJ, Behr J, Brown KK, Colby TV, Cordier JF, Flaherty KR, Lasky JA, Lynch DA, Ryu JH, Swigris JJ, Wells AU, Ancochea J, Bouros D, Carvalho C, Costabel U, Ebina M, Hansell DM, Johkoh T, Kim DS, King TE Jr, Kondoh Y, Myers J, Muller NL, Nicholson AG, Richeldi L, Selman M, Dudden RF, Griss BS, Protzko SL, Schunemann HJ; ATS/ERS/JRS/ALAT Committee on Idiopathic Pulmonary Fibrosis. An official ATS/ERS/JRS/ALAT statement: idiopathic pulmonary fibrosis: evidence-based guidelines for diagnosis and management. Am J Respir Crit Care Med. 2011 Mar 15;183(6):788-824. doi: 10.1164/rccm.2009-040GL. PMID 21471066
- [Background] Kreuter M, Polke M, Walsh SLF, Krisam J, Collard HR, Chaudhuri N, Avdeev S, Behr J, Calligaro G, Corte T, Flaherty K, Funke-Chambour M, Kolb M, Kondoh Y, Maher TM, Molina Molina M, Morais A, Moor CC, Morisset J, Pereira C, Quadrelli S, Selman M, Tzouvelekis A, Valenzuela C, Vancheri C, Vicens-Zygmunt V, Walscher J, Wuyts W, Wijsenbeek M, Cottin V, Bendstrup E. Acute exacerbation of idiopathic pulmonary fibrosis: international survey and call for harmonisation. Eur Respir J. 2020 Apr 3;55(4):1901760. doi: 10.1183/13993003.01760-2019. Print 2020 Apr. PMID 32060068
- [Background] Molyneaux PL, Cox MJ, Willis-Owen SA, Mallia P, Russell KE, Russell AM, Murphy E, Johnston SL, Schwartz DA, Wells AU, Cookson WO, Maher TM, Moffatt MF. The role of bacteria in the pathogenesis and progression of idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2014 Oct 15;190(8):906-13. doi: 10.1164/rccm.201403-0541OC. PMID 25184687
- [Background] O'Dwyer DN, Ashley SL, Gurczynski SJ, Xia M, Wilke C, Falkowski NR, Norman KC, Arnold KB, Huffnagle GB, Salisbury ML, Han MK, Flaherty KR, White ES, Martinez FJ, Erb-Downward JR, Murray S, Moore BB, Dickson RP. Lung Microbiota Contribute to Pulmonary Inflammation and Disease Progression in Pulmonary Fibrosis. Am J Respir Crit Care Med. 2019 May 1;199(9):1127-1138. doi: 10.1164/rccm.201809-1650OC. PMID 30789747
- [Background] Cottin V, Cadranel J, Crestani B, Dalphin JC, Delaval P, Israel-Biet D, Kessler R, Reynaud-Gaubert M, Valeyre D, Wallaert B, Bouquillon B, Cordier JF. Management of idiopathic pulmonary fibrosis in France: a survey of 1244 pulmonologists. Respir Med. 2014 Jan;108(1):195-202. doi: 10.1016/j.rmed.2013.11.017. Epub 2013 Dec 3. PMID 24361163
- [Background] Shulgina L, Cahn AP, Chilvers ER, Parfrey H, Clark AB, Wilson EC, Twentyman OP, Davison AG, Curtin JJ, Crawford MB, Wilson AM. Treating idiopathic pulmonary fibrosis with the addition of co-trimoxazole: a randomised controlled trial. Thorax. 2013 Feb;68(2):155-62. doi: 10.1136/thoraxjnl-2012-202403. Epub 2012 Nov 10. PMID 23143842